CLINICAL TRIAL: NCT03820986
Title: A Phase 3 Randomized, Placebo-controlled Trial to Evaluate the Safety and Efficacy of Pembrolizumab (MK-3475) and Lenvatinib (E7080/MK-7902) Versus Pembrolizumab Alone as First-line Intervention in Participants With Advanced Melanoma (LEAP-003)
Brief Title: Safety and Efficacy Study of Pembrolizumab (MK-3475) Combined With Lenvatinib (MK-7902/E7080) as First-line Intervention in Adults With Advance Melanoma (MK-7902-003/E7080-G000-312/LEAP-003)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7902-003; MK-7902-003 (Other: MSD Protocol Number); E7080-G000-312 (Other: Eisai Protocol Number); LEAP-003 (Other: MSD); 2018-002520-16 (EudraCT Number)
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Malignant Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); programmed cell death-ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule daily for up to at least 2 years.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab+Placebo (Active Comparator): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule daily for up to at least 2 years.
  Interventions: Biological: Pembrolizumab; Drug: Placebo for lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenvatinib — Oral capsule
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Pembrolizumab+Lenvatinib
Drug: Placebo for lenvatinib — Oral capsule
  Arms: Pembrolizumab+Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pembrolizumab (MK-3475) combined with lenvatinib (MK-7902/E7080) compared to pembrolizumab alone (with placebo for lenvatinib) as first-line treatment in adults with no prior systemic therapy for their advanced melanoma.

The primary study hypotheses are that: 1) The combination of pembrolizumab and lenvatinib is superior to pembrolizumab and placebo as assessed by Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), and 2) The combination of pembrolizumab and lenvatinib is superior to pembrolizumab and placebo as assessed by Overall Survival (OS). For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

DETAILED DESCRIPTION:
As of 03-April-2023 active participants, investigator, and sponsor personnel or delegate(s) involved in the treatment administration or clinical evaluation of the participants will be unblinded.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed melanoma.
* Has unresectable Stage III or Stage IV melanoma, as per American Joint Committee on Cancer guidelines, not amenable to local therapy.
* Has been untreated for advanced or metastatic disease except as follows:

  1. Proto-oncogene B-Raf (BRAF) V600 mutation-positive melanoma may have received standard of care targeted therapy as first-line therapy for advanced or metastatic disease. Participants that do not have a BRAF V600 mutation but did receive BRAF or BRAF/mitogen-activated extracellular signal-regulated kinase 1/2 Inhibitor (MEKi) therapy are eligible to participate in this study after discussion with the medical monitor.
  2. Prior adjuvant or neoadjuvant therapy, with targeted therapy or immunotherapy (such as anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], anti-programmed cell death 1 [anti-PD-1] therapy or interferon) will only be permitted if relapse did not occur during active treatment or within 6 months of treatment discontinuation.
* Have documentation of BRAF V600-activating mutation status or consent to BRAF V600 mutation testing during the Screening period (participants with BRAF mutation-positive melanoma as well as BRAF wild-type or unknown are eligible).
* Has an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Has the presence of ≥1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1.
* Provides a tumor biopsy. Participants must submit tumor sample during Screening for confirmation of adequacy of tumor tissue at a central pathology laboratory. Participants who do not submit a tumor tissue sample will not be randomized. The tumor biopsy may not be obtained from a lone target lesion. Confirmation of presence of tumor tissue is not required prior to randomization.
* Has resolution of toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia). If participant received major surgery or radiation therapy of >30 Gray (Gy), they must have recovered from the toxicity and/or complications from the intervention.
* Male participants must agree to use contraception during the treatment period and for at least 7 days after the last dose of study treatment and refrain from donating sperm during this period. Please note that 7 days after lenvatinib/placebo is stopped, if the participant is on pembrolizumab only, no male contraception measures are needed. Contraception use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions is more stringent than the requirements above, the local label requirements are to be followed.
* Female participants must not be pregnant, not breastfeeding, and ≥1 of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP). OR
  2. A WOCBP who agrees to use study-approved contraception during the treatment period and for at least 120 days after the last dose of study treatment.
* The participant (or legally acceptable representative) has provided documented informed consent for the study.
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mmHg at screening and no change in antihypertensive medications within 1 week before Cycle 1 Day 1.
* Has adequate organ function.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early stage cancers (carcinoma in situ or Stage 1, non-ulcerated primary melanoma <1 mm in depth with no nodal involvement) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has ocular melanoma.
* Has known hypersensitivity to active substances or any of their excipients including previous clinically significant hypersensitivity reaction to treatment with another monoclonal antibody.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy.
* Has known history of human immunodeficiency virus (HIV) infection
* Has known history of or is positive for hepatitis B virus or hepatitis C virus infection.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has a history of active tuberculosis (Bacillus tuberculosis).
* Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib.
* Has had a major surgery within 3 weeks prior to first dose of study intervention. Note: Adequate wound healing after major surgery must be assessed clinically independent of time elapsed for eligibility.
* Has a preexisting Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
* Has radiographic evidence of encasement or invasion of major blood vessel, or of intratumoral cavitation.
* Has active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study treatment.
* Has clinically significant cardiovascular disease from 12 months of the first dose of study treatment including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.
* Has urine protein ≥1 g/24-hour. Note: Participants with ≥2+ (≥100 mg/dL) proteinuria on urine dipstick testing (or urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria.
* Prolongation of QTcF interval to >480 ms. Note: If the QTcF is prolonged to >480 ms in the presence of a pacemaker, contact the Sponsor to determine eligibility.
* Has left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range, as determined by multigated acquisition scan (MUGA) or echocardiogram.
* Has received prior therapy in the adjuvant setting. Note: Targeted therapy, anti-CTLA-4, or anti-PD-1 may be allowed.
* Has received prior systemic treatment for unresectable or metastatic melanoma other than targeted therapy as noted in Inclusion Criteria above
* Has received prior therapy with a monoclonal antibody, chemotherapy, or an investigational agent or device within 4 weeks or 5 half-lives (whichever is longer) before administration of study treatment or not recovered (≤Grade 1 or at Baseline) from adverse events due to previously administered agents.

Exception to this rule would be use of denosumab, which is not excluded. Note: Participants with alopecia and ≤Grade 2 neuropathy are an exception and may enroll.

* Has received prior radiotherapy within 2 weeks of first dose of study treatment (Cycle 1 Day 1). Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has received live vaccine within 30 days before the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has had an allogeneic tissue/solid organ transplant.
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (119):
- United States (17):
  - The Angeles Clinic and Research Institute ( Site 0707), Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center ( Site 0704), San Francisco, California
  - California Pacific Medical Center Research Institute ( Site 0705), San Francisco, California
  - John Wayne Cancer Institute ( Site 0706), Santa Monica, California
  - University of Colorado Cancer Center ( Site 0708), Aurora, Colorado
  - Yale Cancer Center ( Site 0709), New Haven, Connecticut
  - Baptist MD Anderson Cancer Center ( Site 0767), Jacksonville, Florida
  - Mid-Florida Cancer Centers ( Site 0764), Orange City, Florida
  - AMG Oncology ( Site 0714), Park Ridge, Illinois
  - Illinois Cancer Care, PC ( Site 0765), Peoria, Illinois
  - Minnesota Oncology Specialist, PA ( Site 0766), Fridley, Minnesota
  - St. Vincent Frontier Cancer Center ( Site 0724), Billings, Montana
  - Atlantic Health System ( Site 0768), Morristown, New Jersey
  - Valley Hospital ( Site 0749), Paramus, New Jersey
  - University of North Carolina - Cancer Hospital ( Site 0751), Chapel Hill, North Carolina
  - OHSU Center for Health & Healing ( Site 0731), Portland, Oregon
  - Inova Schar Cancer Institute ( Site 0739), Fairfax, Virginia
- Australia (6):
  - Lismore Base Hospital ( Site 0453), Lismore, Australian Capital Territory
  - Melanoma Institute Australia ( Site 0452), North Sydney, New South Wales
  - Westmead Hospital ( Site 0451), Westmead, New South Wales
  - Princess Alexandra Hospital ( Site 0454), Wooloongabba, Queensland
  - Eastern Health ( Site 0457), Box Hill, Victoria
  - Fiona Stanley Hospital ( Site 0456), Murdoch, Western Australia
- Austria (2):
  - LKH Universitatsklinikum Graz ( Site 0776), Graz, Styria
  - Medizinische Universitat Wien ( Site 0778), Vienna
- Brazil (5):
  - PERSONAL - Oncologia de Precisao e Personalizada ( Site 0399), Belo Horizonte, Minas Gerais
  - Hospital de Caridade de Ijui ( Site 0391), Ijuí, Rio Grande do Sul
  - Hospital Sao Vicente de Paulo ( Site 0396), Passo Fundo, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 0397), Porto Alegre, Rio Grande do Sul
  - Instituto Nacional de Cancer Hospital do Cancer II ( Site 0394), Rio de Janeiro
- Canada (5):
  - BC Cancer-Kelowna - Sindi Ahluwalia Hawkins Centre ( Site 0661), Kelowna, British Columbia
  - Lions Gate Hospital ( Site 0662), North Vancouver, British Columbia
  - Sunnybrook Research Institute ( Site 0654), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0652), Montreal, Quebec
  - McGill University Health Centre ( Site 0651), Montreal, Quebec
- Chile (5):
  - Fundacion Arturo Lopez Perez FALP ( Site 0421), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0422), Santiago, Region M. de Santiago
  - Sociedad Medica Aren y Bachero Limitada ( Site 0426), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0425), Temuco, Región de la Araucanía
  - Oncocentro ( Site 0424), Viña del Mar, Región de Valparaíso
- China (11):
  - Beijing Cancer Hospital ( Site 0601), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0612), Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 0602), Guangzhou, Guangdong
  - Henan Cancer Hospital ( Site 0610), Zhengzhou, Henan
  - Nanjing Drum Tower Hospital ( Site 0609), Nanjing, Jiangsu
  - The First Hospital Of Jilin University ( Site 0603), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 0607), Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0606), Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital ( Site 0604), Kunming, Yunnan
  - Sir Run Run Shaw Hospital ( Site 0605), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0608), Hangzhou, Zhejiang
- France (10):
  - Hopital ARCHET 2 ( Site 0009), Nice, Alpes-Maritimes
  - Hopital La Timone ( Site 0002), Marseille, Bouches-du-Rhone
  - CHU Dijon Bourgogne ( Site 0010), Dijon, Cote-d Or
  - Institut Claudius Regaud IUCT Oncopole ( Site 0003), Toulouse, Haute-Garonne
  - Hopital Ambroise Pare Boulogne ( Site 0007), Boulogne-Billancourt, Hauts-de-Seine
  - CHRU Lille - Hopital Claude Huriez ( Site 0004), Lille, Nord
  - CHU de Rouen ( Site 0013), Rouen, Seine-Maritime
  - Centre Hospitalier Victor Dupouy ( Site 0012), Argenteuil, Val-d Oise
  - Institut Gustave Roussy ( Site 0001), Villejuif, Val-de-Marne
  - CHU de la Miletrie Poitiers ( Site 0011), Poitiers, Vienne
- Germany (8):
  - Klinik fur Dermatologie Allergologie und Venerologie ( Site 0035), Hannover, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen ( Site 0044), Erlangen, Bavaria
  - Universitaetsklinikum Wuerzburg-Department of Dermatology ( Site 0036), Würzburg, Bavaria
  - Hautkrebszentrum Buxtehude ( Site 0037), Buxtehude, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus ( Site 0041), Dresden, Saxony
  - Universitaetsklinikum Leipzig ( Site 0040), Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel ( Site 0033), Kiel, Schleswig-Holstein
  - SRH Wald-Klinikum Gera GmbH ( Site 0042), Gera, Thuringia
- Israel (8):
  - HaEmek Medical Center ( Site 0306), Afula
  - Soroka Medical Center ( Site 0303), Beersheba
  - Rambam Medical Center ( Site 0301), Haifa
  - Hadassah Ein Karem Hebrew University Medical Center ( Site 0305), Jerusalem
  - Rabin Medical Center ( Site 0302), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0304), Ramat Gan
  - Sourasky Medical Center ( Site 0307), Tel Aviv
  - Shamir Medical Center-Assaf Harofeh ( Site 0308), Ẕerifin
- Italy (6):
  - ASST Papa Giovanni XXIII ( Site 0062), Bergamo, Abruzzo
  - Azienda Ospedaliera Universitaria Senese ( Site 0065), Siena, Tuscany
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0064), Milan
  - Istituto Europeo di Oncologia ( Site 0067), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 0061), Napoli
  - Istituto Oncologico Veneto ( Site 0063), Padua
- Poland (5):
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwers Medyczn ( Site 0272), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im.prof. F. Lukaszczyka w Bydgoszczy ( Site 0273), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow ( Site 0280), Krakow, Lesser Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0281), Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 0278), Gliwice, Silesian Voivodeship
- South Africa (3):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 0805), Port Elizabeth, Eastern Cape
  - Sandton Oncology Medical Group PTY LTD ( Site 0802), Johannesburg, Gauteng
  - Cape Town Oncology Trials Pty Ltd ( Site 0803), Kraaifontein, Western Cape
- South Korea (4):
  - Kyungpook National University Chilgok Hospital ( Site 0553), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 0554), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0552), Seoul
  - Samsung Medical Center ( Site 0551), Seoul
- Spain (9):
  - Hospital Duran i Reinals ICO de Hospitalet ( Site 0187), Hospitalet Del Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla ( Site 0181), Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruna. CHUAC ( Site 0182), A Coruña, La Coruna
  - Hospital Universitario Insular de Gran Canaria ( Site 0189), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Clinic i Provincial Barcelona ( Site 0190), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 0191), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 0183), Madrid
  - Hospital Universitario La Paz ( Site 0184), Madrid
  - Hospital Universitario Carlos Haya ( Site 0186), Málaga
- Sweden (7):
  - Laenssjukhuset Ryhov ( Site 0215), Jönköping, Jönköping County
  - Centrallasarettet Vaxjo ( Site 0214), Vaxjo, Kronoberg County
  - Skanes Universitetssjukhus ( Site 0213), Lund, Skåne County
  - Karolinska Universitetssjukhuset ( Site 0211), Solna, Stockholm County
  - Akademiska Sjukhuset ( Site 0218), Uppsala, Uppsala County
  - Norrlands Universitetssjukhus ( Site 0216), Umeå, Västerbotten County
  - Sahlgrenska Universitetssjukhuset ( Site 0212), Gothenburg, Västra Götaland County
- Switzerland (4):
  - Universitaetsspital Basel ( Site 0094), Basel, Canton of Basel-City
  - Kantonsspital Winterthur ( Site 0095), Winterthur, Canton of Zurich
  - Universitaetsspital Zuerich ( Site 0092), Zuerich-Flughafen, Canton of Zurich
  - Kantonsspital Graubuenden ( Site 0091), Chur, Kanton Graubünden
- United Kingdom (4):
  - Western General Hospital ( Site 0121), Edinburgh, Edinburgh, City of
  - Guys and St Thomas NHS Foundation Trust ( Site 0126), London, London, City of
  - Derriford Hospital ( Site 0129), Plymouth
  - Singleton Hospital ( Site 0131), Swansea

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Arance A, Berciano-Guerrero MA, Guo J, Carlino MS, Ascierto PA, Burotto M, Mortier L, Queirolo P, Chiarion-Sileni V, Schachter J, Zhang X, Martin-Liberal J, Del Vecchio M, Okpara CE, Dutcus C, Zhang J, Diede SJ, Neff T, Long GV. Randomized, double-blind, phase III LEAP-003 study of first-line lenvatinib plus pembrolizumab versus placebo plus pembrolizumab for unresectable or metastatic melanoma. Ann Oncol. 2025 Dec;36(12):1535-1546. doi: 10.1016/j.annonc.2025.08.008. Epub 2025 Aug 28. PMID 40885529
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26976&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adult participants with advanced melanoma, who have not received prior systemic therapy were enrolled. 674 participants were randomly assigned in a 1:1 ratio to either combination therapy, Pembrolizumab+Lenvatinib, or Pembrolizumab+Placebo, to assess the safety and efficacy of combination therapy, Pembrolizumab+Lenvatinib.
Groups:
- Pembrolizumab+Lenvatinib: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule daily for up to at least 2 years.
- Pembrolizumab+Placebo: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule daily for up to at least 2 years.
Period: Overall Study
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Started | 334 | 340
Treated | 332 | 338
Completed | 0 | 0
Not Completed | 334 | 340
Not completed — Death | 201 | 175
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Decision | 122 | 160
Not completed — Withdrawal by Subject | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo | Total
Number analyzed (Participants) | 334 | 340 | 674
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (14.0) | 62.0 (13.1) | 61.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 139 | 264
  Male | 209 | 201 | 410
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 79 | 149
  Not Hispanic or Latino | 224 | 225 | 449
  Unknown or Not Reported | 40 | 36 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 55 | 43 | 98
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 243 | 261 | 504
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 34 | 31 | 65
Proto-oncogene B-Raf (BRAF) mutation positive [Count of Participants; unit: Participants] — Participants were stratified according to BRAF mutation status: BRAF mutation-positive, or BRAF wild-type or unknown.
  Participants
    No | 211 | 215 | 426
    Yes | 123 | 125 | 248

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) Per Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 34 months
Population: All randomized participants, included in the treatment group to which they were randomized. The final analysis for this outcome is presented here.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 334 | 340
Months | 9.1 [6.4 to 11.8] | 4.2 [3.1 to 6.3]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Test type: Superiority — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate and stratified by BRAF mutation positive (Yes vs. No); p = 0.0176, Log Rank; One-sided p-value based on log-rank test and stratified by BRAF mutation positive (Yes vs. No); Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.67 to 0.98] — HR=Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to date of death from any cause. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 46 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 334 | 340
Months | 25.8 [23.0 to 33.9] | 39.5 [26.6 to NA] — NA=upper limit not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Test type: Superiority — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate and stratified by BRAF mutation positive (Yes vs. No); p = 0.9521, Log Rank; One-sided p-value based on log-rank test and stratified by BRAF mutation positive (Yes vs. No); Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.97 to 1.48] — HR=Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by BICR Per RECIST 1.1
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 46 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 334 | 340
Percentage of participants | 43.4 [38.0 to 48.9] | 35.6 [30.5 to 40.9]

4. Secondary Outcome: Duration of Response (DOR) as Assessed by BICR Per RECIST 1.1
Description: For participants who demonstrated CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the date of the first documented evidence of CR or PR until disease progression or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. For this study, RECIST 1.1 has been modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 46 months
Population: Randomized participants who had a confirmed complete or partial response, included in the treatment group to which they were randomized. The final analysis for this outcome is presented here.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 145 | 121
Months | 26.9 [3.4 to NA] — NA=upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event.

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 67 months
Population: All randomized participants who received at least one dose of study intervention. The final analysis for this outcome is presented here.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 332 | 338
Participants | 331 | 330

6. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued any study treatment due to an AE is presented. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 63 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 332 | 338
Participants | 104 | 68

7. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire-Core 30 [QLQ-C30] Global Health Status (GHS)/Quality of Life (QoL) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The GHS/QoL combined score consists of participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" GHS/QoL responses range in score from 0 to 100, with a higher score indicating a better outcome. The final analysis for this outcome is presented here.
Time Frame: Baseline and Week 21
Population: All randomized participants who had at least 1 assessment available for the EORTC QLQ-C30 GHS/QoL score and had received at least 1 dose of study intervention. The final analysis for this outcome is presented here.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 325 | 334
Scores on a scale | -6.38 [-8.91 to -3.84] | -2.69 [-5.30 to -0.08]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Based on a constrained longitudinal data analysis (cLDA) model with GHS/QoL as the response variable, with covariates for treatment by time interaction, stratification factor BRAF mutation status as covariate. No formal hypothesis testing was conducted. P-value is nominal; Test type: Other; p = 0.0345, cLDA model — No formal hypothesis testing was conducted. P-value is nominal; Difference in LS means = -3.69, 95% CI 2-sided [-7.10 to -0.27] — Difference in LS means=Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire-Core 30 [QLQ-C30] Physical Function (PF) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The PF Score consists of participant responses to questions regarding PF (5 questions about daily activities [strenuous activities, long walks, short walks, bed/chair rest and needing help with eating, dressing, washing themselves or using the toilet]). For PF, responses range in score from 0 to 100, with a higher score indicating a better outcome. The final analysis for this outcome is presented here.
Time Frame: Baseline and Week 21
Population: All randomized participants who had at least 1 assessment available for the EORTC QLQ-C30 PF score and had received at least 1 dose of study intervention. The final analysis for this outcome is presented here.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 325 | 334
Scores on a scale | -9.50 [-11.66 to -7.34] | -4.02 [-6.23 to -1.80]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Based on a cLDA model with PF as the response variable, with covariates for treatment by time interaction, stratification factor BRAF mutation status as covariate. No formal hypothesis testing was conducted. P-value is nominal; Test type: Other; p = 0.0004, cLDA model; No formal hypothesis testing was conducted. P-value is nominal; Difference in LS means = -5.49, 95% CI 2-sided [-8.53 to -2.45] — Difference in LS means=Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo

9. Secondary Outcome: Time to True Deterioration (TTD) Based on Change From Baseline in EORTC QLQ-C30 GHS/QoL Score
Description: TTD is defined as the time from Baseline to 1st onset of a ≥10-point negative change (decrease) in EORTC-QLQ-C30 GHS Score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The GHS/QoL Score consists of participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" GHS/QoL responses range in score from 0 to 100, with a higher score indicating a better outcome. A longer TTD indicates a better outcome. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 30 months
Population: Per protocol, the analysis population consisted of all randomized participants who have at least one assessment available for EORTC QLQ-C30 and have received at least one dose of the study intervention; and had data available for this TTD change from baseline in GHS/QoL outcome using EORTC QLQ-C30. The final analysis for this outcome is presented here.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 305 | 323
Months | 5.62 [4.34 to 9.69] | 24.58 [11.04 to NA] — NA=not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by BRAF mutation status (positive vs wild type or unknown) No formal hypothesis testing was conducted. P-value is nominal; Test type: Other; p = 0.0001, Log Rank; No formal hypothesis testing was conducted. P-value is nominal; Hazard Ratio (HR) = 1.58, 95% CI 2-sided [1.25 to 2.00] — HR=Lenvatinib + Pembrolizumab vs. Placebo + Pembrolizumab

10. Secondary Outcome: Time to True Deterioration (TTD) Based on Change From Baseline in EORTC QLQ-C30 in Physical Function (PF) Score
Description: TTD is defined as the time from Baseline to 1st onset of a ≥10-point negative change (decrease) in EORTC-QLQ-C30 PF Score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The PF Score consists of participant responses to questions regarding PF (5 questions about daily activities [strenuous activities, long walks, short walks, bed/chair rest & needing help with eating, dressing, washing themselves or using the toilet]. For PF, responses range in score from 0 to 100, with a higher score indicating a better outcome. The final analysis for this outcome is presented here.
Time Frame: Up to approximately 30 months
Population: Per protocol, the analysis population consisted of all randomized participants who have at least one assessment available for EORTC QLQ-C30 and have received at least one dose of the study intervention; and had data available for this TTD change from baseline in PF Score outcome using EORTC QLQ-C30. The final analysis for this outcome is presented here.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
Number analyzed (Participants) | 305 | 323
Months | 5.55 [4.40 to 9.69] | NA [NA to NA] — NA=not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Pembrolizumab+Placebo; Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by BRAF mutation status (positive vs wild type or unknown). No formal hypothesis testing was conducted. P-value is nominal; Test type: Other; p = .0001, Log Rank; No formal hypothesis testing was conducted. P-value is nominal; Hazard Ratio (HR) = 1.95, 95% CI 2-sided [1.52 to 2.50] — HR=Lenvatinib + Pembrolizumab vs. Placebo + Pembrolizumab

ADVERSE EVENTS:
Time Frame: Up to approximately 67 months
Description: All-cause mortality includes all randomized participants included into treatment group they were randomized. Serious AEs & other AEs: includes all randomized participants who received ≥1 dose of study intervention. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab+Lenvatinib | Pembrolizumab+Placebo
All-Cause Mortality (participants affected / at risk) | 206/334 | 176/340
Serious Adverse Events (participants affected / at risk) | 124/332 | 96/338
Other Adverse Events (participants affected / at risk) | 326/332 | 319/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Lenvatinib (N=332) | Pembrolizumab+Placebo (N=338)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (4) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 6 (6)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Tick-borne fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (6)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 3 (3)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 3 (4) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Lenvatinib (N=332) | Pembrolizumab+Placebo (N=338)
Anaemia (Blood and lymphatic system disorders) | 40 (58) | 53 (70)
Neutropenia (Blood and lymphatic system disorders) | 25 (43) | 8 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (32) | 6 (6)
Hyperthyroidism (Endocrine disorders) | 44 (48) | 17 (18)
Hypothyroidism (Endocrine disorders) | 157 (198) | 44 (50)
Abdominal pain (Gastrointestinal disorders) | 58 (96) | 40 (45)
Abdominal pain upper (Gastrointestinal disorders) | 47 (58) | 19 (22)
Constipation (Gastrointestinal disorders) | 59 (90) | 50 (60)
Diarrhoea (Gastrointestinal disorders) | 171 (454) | 84 (141)
Dry mouth (Gastrointestinal disorders) | 36 (39) | 23 (26)
Dyspepsia (Gastrointestinal disorders) | 31 (39) | 12 (13)
Nausea (Gastrointestinal disorders) | 111 (204) | 61 (85)
Stomatitis (Gastrointestinal disorders) | 30 (43) | 4 (4)
Vomiting (Gastrointestinal disorders) | 75 (134) | 38 (51)
Asthenia (General disorders) | 95 (164) | 82 (122)
Fatigue (General disorders) | 92 (130) | 86 (109)
Mucosal inflammation (General disorders) | 39 (54) | 10 (12)
Oedema peripheral (General disorders) | 39 (43) | 34 (43)
Pyrexia (General disorders) | 40 (50) | 42 (60)
COVID-19 (Infections and infestations) | 21 (21) | 28 (33)
Urinary tract infection (Infections and infestations) | 28 (39) | 35 (44)
Alanine aminotransferase increased (Investigations) | 75 (118) | 55 (89)
Amylase increased (Investigations) | 47 (73) | 37 (72)
Aspartate aminotransferase increased (Investigations) | 82 (130) | 47 (67)
Blood alkaline phosphatase increased (Investigations) | 34 (52) | 24 (30)
Blood bilirubin increased (Investigations) | 40 (81) | 19 (34)
Blood cholesterol increased (Investigations) | 36 (77) | 13 (27)
Blood creatine phosphokinase increased (Investigations) | 49 (77) | 41 (73)
Blood creatinine increased (Investigations) | 42 (73) | 26 (48)
Blood glucose increased (Investigations) | 18 (40) | 16 (28)
Blood lactate dehydrogenase increased (Investigations) | 33 (63) | 21 (28)
Blood sodium decreased (Investigations) | 21 (46) | 10 (19)
Blood thyroid stimulating hormone increased (Investigations) | 56 (79) | 18 (36)
Blood triglycerides increased (Investigations) | 31 (67) | 22 (43)
Blood urea increased (Investigations) | 21 (38) | 14 (43)
Gamma-glutamyltransferase increased (Investigations) | 36 (49) | 23 (30)
Lipase increased (Investigations) | 85 (171) | 61 (115)
Platelet count decreased (Investigations) | 26 (42) | 3 (3)
Weight decreased (Investigations) | 91 (111) | 30 (36)
Decreased appetite (Metabolism and nutrition disorders) | 113 (166) | 54 (58)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 35 (64) | 18 (27)
Hyperglycaemia (Metabolism and nutrition disorders) | 52 (92) | 39 (62)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 59 (118) | 28 (49)
Hyperuricaemia (Metabolism and nutrition disorders) | 17 (29) | 9 (16)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (33) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 37 (51) | 16 (23)
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 (27) | 9 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 37 (57) | 20 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 100 (162) | 69 (100)
Back pain (Musculoskeletal and connective tissue disorders) | 64 (78) | 42 (56)
Myalgia (Musculoskeletal and connective tissue disorders) | 63 (76) | 42 (52)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 (37) | 32 (38)
Dizziness (Nervous system disorders) | 40 (54) | 27 (29)
Dysgeusia (Nervous system disorders) | 23 (32) | 5 (6)
Headache (Nervous system disorders) | 76 (131) | 51 (59)
Insomnia (Psychiatric disorders) | 25 (29) | 29 (30)
Proteinuria (Renal and urinary disorders) | 100 (177) | 35 (61)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (51) | 41 (54)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 54 (61) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (30) | 25 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (22) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (23) | 12 (12)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 52 (71) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 68 (81) | 78 (114)
Rash (Skin and subcutaneous tissue disorders) | 62 (89) | 57 (75)
Vitiligo (Skin and subcutaneous tissue disorders) | 21 (23) | 41 (41)
Hypertension (Vascular disorders) | 203 (378) | 75 (119)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03820986/Prot_SAP_001.pdf